CLINICAL TRIAL: NCT01791764
Title: Hospital Mortality After ST Segment Elevation Acute Myocardial Infarction Submitted to Pharmacoinvasive Strategy With Tenecteplase (TNK): Analysis of 398 Patients.
Brief Title: Hospital Mortality in Patients Submitted to Pharmacoinvasive Strategy With Tenecteplase (TNK)
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Felipe José de Andrade Falcão, Master, Federal University of São Paulo
Other Study IDs: SAMU-01
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study has the following objective:

To identify related factors to hospital mortality in patients with ST-segment elevation acute myocardial infarction submitted to pharmacoinvasive strategy within a structured healthcare network.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention is the main therapy for patients with ST-segment elevation acute myocardial infarction. However, a significant portion of these patients won't receive optimal treatment due to the small number of tertiary centers with interventional laboratories available for 24 hours a day, 7 days a week.

Specially in large urban centers and rural areas, where tertiary care hospitals are restricted to a specific region, alternative approaches must be developed. The pharmacoinvasive strategy has emerged as an alternative for patients admitted to primary care centers. It is based in up-front intravenous thrombolytic therapy and transfer to a tertiary center where early, systematic, coronary intervention will be performed between 3 to 24 hours after the administration of thrombolytic drugs, even in cases in which successful reperfusion was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ST-segment elevation acute myocardial infarction submitted to pharmacoinvasive strategy with tenecteplase.

Exclusion Criteria:

* Absence of obstructive coronary disease
* Surgical reference
* Did not undergo catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | During hospital stay,an expected average of 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Felipe JA Falcao, Principal Investigator — Federal University of São Paulo; Claudia MR Alves, Doctor, Principal Investigator — Federal University of São Paulo; Antonio CC Carvalho, Study Director — Federal University of São Paulo; Adriano HP Barbosa, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Falcao FJ, Alves CM, Barbosa AH, Caixeta A, Sousa JM, Souza JA, Amaral A, Wilke LC, Perez FC, Goncalves Junior I, Stefanini E, Carvalho AC. Predictors of in-hospital mortality in patients with ST-segment elevation myocardial infarction undergoing pharmacoinvasive treatment. Clinics (Sao Paulo). 2013 Dec;68(12):1516-20. doi: 10.6061/clinics/2013(12)07. PMID 24473509